CLINICAL TRIAL: NCT06497166
Title: Examining of Occupational Balance, Executive Functions, and Quality of Life of Adolescents Diagnosed with Internet Gaming Disorder
Brief Title: Examining of Occupational Balance, Executive Functions, and Quality of Life of Adolescents with Internet Gaming Disorder
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Beyzanur Demirci, Research Assistant, Bezmialem Vakif University
Other Study IDs: BEZMIALEM-BDEMIRCI-2024-001
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Internet Addiction Disorder
Keywords: Addiction; Executive functions; Internet gaming disorder; Occupational balance; Quality of life
MeSH Terms: conditions — Internet Addiction Disorder; Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Research Group: 12-18 year old adolescents diagnosed with internet gaming disorder
- Control Group: 12-18 year old healthy adolescents

SUMMARY:
Internet gaming disorder leads to social problems and isolation, neglect of daily responsibilities, behavioral disorders, and cognitive and physical impairments. It is thought that assessing the occupational profiles and cognitive functions of adolescents with internet gaming disorder will bring a new perspective to the occupational therapy literature. The aim of the present study is to examine the occupational balance, executive functions, and quality of life of adolescents with internet gaming disorder.

DETAILED DESCRIPTION:
The study, planned to be conducted with individuals aged 12-18 who are followed up in the Child and Adolescent Mental Health and Diseases outpatient clinic of Bezmialem Vakif University and diagnosed with internet gaming disorder according to DSM-V diagnostic criteria, will include a total of 62 participants, with 31 in the study group and 31 in the healthy control group. All individuals who provide written consent will be administered the Sociodemographic Data Form, Internet Gaming Disorder Scale, Teenage Executive Function Inventory, Pediatric Quality of Life Inventory-Adolescent Form, and Adolescent Occupational Balance Scale, and the results will be recorded. The obtained results will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Internet Gaming Disorder
* Aged between 12 and 18
* Proficiency in Turkish
* Open to communication and cooperation
* Willing to participate in the study
* No reported cognitive impairment

Exclusion Criteria:

* Additional psychiatric diagnosis
* Having a neurological problem that would impair communication and collaboration

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents diagnosed with internet gaming disorder
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Adolescent Occupational Balance Scale | Baseline
  The scale measures occupational balance. According to the four-point Likert rating, the lowest raw score to be taken from the scale is 27, and the highest raw score is 108. It takes approximately 15-20 min to respond to the whole scale. A high score obtained from the scale indicates a high level of occupational balance.
Teenage Executive Functioning Inventory | Baseline
  The scale measures executive functioning. It is a 5-point Likert type inventory and includes statements scored from 1 to 5 (1: Definitely not true, 5: Definitely true). Higher scores represent more difficulty with executive functions. The lowest score to be taken from the scale is 20, and the highest score is 100.
Pediatric Quality of Life Inventory | Baseline
  The scale measures quality of life. It is a 23-item measurement tool. Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3= 25, 4 = 0), so that higher scores indicate better quality of life. This instrument yields a Total score, Physical Health Summary score (Equivalent to the Physical Functioning subscale) and Psychosocial Health Summary score (Based on the Emotional Functioning subscale, Social Functioning subscale, and School Functioning subscale). The lowest score to be taken from the scale is 0, and the highest score is 100.
Internet Gaming Disorder Scale | Baseline
  The scale measures internet gaming disorder severity. The lowest score that can be obtained from the scale is 20 and the highest score is 100. Higher scores indicate a more severe disorder.
Sociodemographic Information Form | Baseline
  Measures sociodemographic information

CONTACTS AND LOCATIONS:
Overall Officials: Beyzanur Demirci, MSc, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided